CLINICAL TRIAL: NCT03856437
Title: A Message Framing Intervention for Increasing Parental Acceptance of Human Papillomavirus Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1322177-1.1; R01CA219060 (NIH)
Record Dates: First submitted 2018-12-17; First posted 2019-02-27 (Actual); Results first posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Cervical Cancer; Anal Cancer; Penile Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Anus Neoplasms; Penile Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gain-framed messages (Experimental): Participants in this arm receive gain-framed HPV vaccination messages.
  Interventions: Behavioral: HPV vaccination messages
- Loss-framed messages (Experimental): Participants in this arm receive loss-framed HPV vaccination messages.
  Interventions: Behavioral: HPV vaccination messages
- Control messages (Active Comparator): Participants in this arm receive non-framed HPV vaccination messages.
  Interventions: Behavioral: HPV vaccination messages

INTERVENTIONS:
Behavioral: HPV vaccination messages — Digital multimedia messages consisting of text and imagery conveying the benefits of being vaccinated against HPV, the costs of not being vaccinated against HPV, or neither benefits or costs but simply a call for action.

SUMMARY:
The goal of this study is to determine the effects of message framing (gain vs. loss) on African American parents' acceptance of the HPV vaccine and how such effects are moderated by parents' salient beliefs prior to message exposure. Participants are randomized into gain and loss conditions in which they view either gain-framed or loss-framed HPV vaccination messages. Key outcome variables include parents' attitudes and intentions toward vaccinating their children against HPV.

DETAILED DESCRIPTION:
The goal of this study is to determine the effects of message framing (gain vs. loss) on African American parents' acceptance of the HPV vaccine and how such effects are moderated by parents' salient beliefs prior to message exposure. Participants recruited from local communities and online panels will complete a computer-assisted survey. In the survey participants will first answer questions related to their beliefs about HPV and the HPV vaccine (e.g., perceived susceptibility, perceived severity, perceived efficacy, perceived safety, etc.), as well as other background information. Then they will be presented with either a gain-framed or loss-framed human papillomavirus vaccination message. After the message exposure, they will answer questions related to their attitudes toward HPV vaccination, intentions to vaccinate their children, as well as other message response measures. Eligible participants are at least 21 years old, self-identify as African American, and are custodial parents or caretakers of at least one child ages 9-17 who has not initiated the HPV vaccine series.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Self-identify as African American
* Custodial parent or caretaker of at least one child under the age of 18 who has not been fully vaccinated against HPV.
* Has access to Internet to complete the study

Exclusion Criteria:

* Younger than 18 years
* Does not self-identify as African American
* Not a custodial parent or caretaker of at least one child under the age of 18 who has not been fully vaccinated against HPV.
* Has no access to Internet to complete the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1170 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2022-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Nan, Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Maryland, College Park, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gain-framed Messages | Loss-framed Messages | Control Messages
Started | 380 | 407 | 383
Completed | 380 | 407 | 383
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gain-framed Messages | Loss-framed Messages | Control Messages | Total
Number analyzed (Participants) | 380 | 407 | 383 | 1170
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.10 (8.59) | 38.64 (8.86) | 38.05 (8.81) | 38.27 (8.75)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 103 | 99 | 111 | 313
  Female | 272 | 299 | 262 | 833
  Non-Binary | 3 | 5 | 5 | 13
  Other | 2 | 4 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 380 | 407 | 383 | 1170
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Baseline Attitudes [Mean (Standard Deviation); unit: units on a scale] — Baseline attitudes toward HPV vaccination for children Scale range: 1-7 (higher score indicates more positive attitude) Subscales were averaged.
  units on a scale | 5.35 (1.77) | 5.30 (1.93) | 5.37 (1.87) | 5.34 (1.86)

OUTCOME MEASURES:

1. Primary Outcome: Attitudes
Description: Attitudes toward HPV vaccination for children Scale range: 1-7 (higher score indicates more positive attitude) Subscales were averaged.
Time Frame: baseline posttest (test was approximately 5 minutes to complete)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gain-framed Messages | Loss-framed Messages | Control Messages
Number analyzed (Participants) | 380 | 407 | 383
score on a scale | 5.61 (1.74) | 5.56 (1.94) | 5.51 (1.87)

2. Primary Outcome: Intention to Vaccinate Free of Cost
Description: Intention to have children vaccinated against HPV free of cost Scale range: 1-6 (higher score indicates stronger intention) Subscales were averaged.
Time Frame: baseline posttest (test was approximately 5 minutes to complete)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gain-framed Messages | Loss-framed Messages | Control Messages
Number analyzed (Participants) | 380 | 407 | 383
units on a scale | 4.56 (1.57) | 4.59 (1.64) | 4.46 (1.70)

3. Secondary Outcome: Intention to Vaccinate With Cost
Description: Intention to have children vaccinated against HPV free with cost Scale range: 1-6 (higher score indicates stronger intention) Subscales were averaged.
Time Frame: baseline posttest (test was approximately 5 minutes to complete)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gain-framed Messages | Loss-framed Messages | Control Messages
Number analyzed (Participants) | 380 | 407 | 383
units on a scale | 4.17 (1.70) | 4.27 (1.79) | 4.08 (1.82)

ADVERSE EVENTS:
Description: Deaths and/or adverse events were not monitored/assessed as this was an online study where participants completed the survey on their own computer at a location of their choice.
Arm/Group | Gain-framed Messages | Loss-framed Messages | Control Messages
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The online survey-experiment may not fully reflect how individuals typically encounter health messages in the real world. There is concern about ecology validity. Also the long-term effects of message exposure were not determined.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/37/NCT03856437/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/37/NCT03856437/SAP_001.pdf
  • Informed Consent Form (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/37/NCT03856437/ICF_002.pdf